CLINICAL TRIAL: NCT04833075
Title: Real World Pharmacokinetics of Immune Checkpoint Inhibitors
Acronym: ELICIT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Approx. half of all samples withdrawn are readily available from another institute. Hence, it is unethical to draw more blood from patients in the ELICIT-trial.
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ELICIT
Record Dates: First submitted 2021-03-30; First posted 2021-04-06 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2022-09

CONDITIONS: Cancer
Keywords: Immune Checkpoint Inhibitor; Pharmacokinetics
MeSH Terms: conditions — Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: A low-interventional cross-sectional pharmacokinetic study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm (Other): additional blood sampling (single arm)
  Interventions: Other: blood sampling

INTERVENTIONS:
Other: blood sampling — A maximum of 13 blood samples (39 mL) will be derived from subjects on treatment. After discontinuation of ICI treatment, a maximum of 7 blood samples (21 mL) will be derived.

SUMMARY:
Rationale: Real-world pharmacokinetic data from cancer patients treated with immune checkpoint inhibitors (ICIs) are sparse. Moreover, pharmacokinetic parameters may be associated with response to ICI treatment and may act as a predictive or early response biomarker.

Objective: To describe the real-world pharmacokinetics of ICIs in patients eligible for ICI treatment or already treated with ICIs.

Study design: A low-interventional cross-sectional pharmacokinetic study. Study population: Patients treated with ICIs. Intervention: A maximum of 13 blood samples (39 mL) will be derived from subjects on treatment. After discontinuation of ICI treatment, a maximum of 7 blood samples (21 mL) will be derived.

Main study parameters: Real- world pharmacokinetic parameters of ICIs: clearance, volume of distribution, serum exposure (serum concentration - time curve).

ELIGIBILITY:
Inclusion Criteria:

* Treatment with immune checkpoint inhibitors (atezolizumab (Tecentriq®), avelumab (Bavencio®), cemiplimab (Libtayo®), durvalumab (Imfinzi®), ipilimumab (Yervoy®), nivolumab (Opdivo®) and pembrolizumab (Keytruda®))
* Willingness and ability to provide written informed consent
* Age 18 years or older

Exclusion Criteria: n/a (real-world)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Real-world pharmacokinetic parameters --> clearance | t=0 until t=12 months or end-of-treatment, whichever comes first (on-treatment) and t=0 until max. t=26 weeks (after discontinuation)(depends on ICI used)
  baseline clearance, change of clearance during treatment
Real-world pharmacokinetic parameters --> volume of distribution | t=0 until t=12 months or end-of-treatment, whichever comes first (on-treatment) and t=0 until max. t=26 weeks (after discontinuation)(depends on ICI used)
  volume of distribution
Real-world pharmacokinetic parameters --> exposure | t=0 until t=12 months or end-of-treatment, whichever comes first (on-treatment) and t=0 until max. t=26 weeks (after discontinuation)(depends on ICI used)
  serum exposure (serum concentration - time curve)

CONTACTS AND LOCATIONS:
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided